CLINICAL TRIAL: NCT04313036
Title: Phase II Open Label Study to Assess Efficacy of 5-day Defibrotide Treatment for Hepatic SOS/VOD
Brief Title: 5-day Defibrotide Treatment for Hepatic SOS/VOD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Hagen, Patrick A, Assistant Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 212665
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Sinusoidal Obstruction Syndrome; Veno-occlusive Disease; Bone Marrow Transplant Complications
Keywords: defibrotide; Sinusoidal; Veno-occlusive; Bone Marrow Transplant; allogeneic stem cell transplant
MeSH Terms: conditions — Hepatic Veno-Occlusive Disease | interventions — defibrotide

STUDY DESIGN:
Intervention Model Description: The goal of this study is to assess the 100-day survival of a 5-day defibrotide treatment for hepatic SOS in allogeneic stem cell transplant patients compared to the standard 21-day treatment. It is hypothesized that the 5-day treatment will have non-inferior 100-day survival rates to the 21-day treatment. Historically, 100-day survival has been 58.9% in moderate and 38.2% in severe SOS. Investigators believe that the null survival for the 21-day defibrotide treatment is 50%. Investigators wish to determine non-inferiority of the 5-day treatment with a 5% margin of error.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Defibrotide (Experimental): 5 day course of defibrotide at standard dosing 25 mg/kg/day in 4 divided doses of 6.25 mg/kg. If not in CR by day 5, will be given for >/= 21 days or per discretion of enrolling physician.
  Interventions: Drug: Defibrotide

INTERVENTIONS:
Drug: Defibrotide — 25 mg/kg/day at 4 divided doses of 6.25 mg/kg, 2-h infusion given for 5 days, if not in CR treatment continued for >/= 21 days or per discretion of enrolling physician.

SUMMARY:
Sinusoidal Obstruction Syndrome (SOS), also referred to as hepatic veno-occlusive disease (VOD), is rare but serious complication of allogeneic stem cell transplantation (allo-SCT). Defibrotide is the only FDA approved therapy to treat SOS and has significantly improved outcomes. When applied early, SOS symptoms often quickly improve and an abbreviated course can be applied. This study is looking at an abbreviated 5 day course of defibrotide in those patients with a complete response to therapy with the primary outcome being day 100 overall survival as compared to history data.

DETAILED DESCRIPTION:
Sinusoidal obstructive syndrome (SOS) has a reported mean incidence of 13.7% and even among those undergoing reduced intensity conditioning regimens is approximately 9%. SOS is a clinical syndrome characterized by painful hepatomegaly, jaundice, ascites, fluid retention, and weight gain. The onset is usually before day 35 after stem cell infusion. SOS ranges in severity from a mild reversible disease to a severe syndrome associated with multiorgan failure (MOF) and death. Prior to the introduction of defibrotide, severe SOS was nearly universally fatal with a mortality rate approaching 100% by day 100 after allo-SCT.

The diagnosis of SOS/VOD is clinical and should be considered in any patient who has undergone hematopoietic stem cell transplantation and develops liver dysfunction. Patients with mild or moderate disease have reasonably good outcomes with supportive therapy alone while in contrast prognosis is much worse in severe SOS which occurs in about 25-30% cases.

Defibrotide is the only established Food and Drug Administration (FDA) approved therapy to treat SOS. It is now approved for use in adults and children with SOS with renal or pulmonary dysfunction following HCT. The standard treatment is 25 mg/kg/day in 4 divided doses of 6.25 mg/kg for 21 days. However, responses are frequently brisk and complete in many patients thus it has been postulated that in responding patients this treatment course could be abbreviated given the risk for adverse events such as hypotension/shock and hemorrhage.

This is an open label pilot study evaluating an abbreviated 5 (as compared to 21) day course of defibrotide in patients with confirmed SOS. The primary outcome is day 100 survival as compared to historical data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent allogeneic stem cell transplantation
2. Age >/= 18 years
3. Diagnosed hepatic SOS/VOD either by Baltimore Criteria or Modified Seattle Criteria including up to 60 days post-transplantation.

Exclusion Criteria:

1. Significant uncontrolled bleeding
2. Prior or concurrent systemic t-PA
3. Concomitant use of therapeutic heparin or other anticoagulants (except use of heparin for central access patency)
4. Hemodynamic instability (>1 pressor gent to maintain blood pressure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-03-11 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Day 100 overall survival | 100 days
  Assess day 100 survival of 5-day defibrotide treatment for hepatic SOS/VOD in allogeneic stem cell transplant patients compared to standard 21-day treatment in the reported literature.

SECONDARY OUTCOMES:
Complete response day 100 | 100 days
  Assess complete response (CR) rates for hepatic SOS/VOD by day +100 defined as resolution of parameters used to document SOS/VOD.
Complete response day 5 | 5 days
  Assess complete response (CR) rates for hepatic SOS/VOD by day +5 as defined by resolution of parameters used to document SOS/VOD.
Complete response day 30 | 30 days
  Assess complete response (CR) rates for hepatic SOS/VOD by day +30 as defined by resolution of parameters used to document SOS/VOD.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick A Hagen, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No